CLINICAL TRIAL: NCT02527369
Title: Effect of the XP1100RF Therapy on Thighs Circumference Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version1-713/2/2014
Record Dates: First submitted 2015-07-30; First posted 2015-08-19 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Thighs Circumferential Reduction; Subcutaneous Fat Cell Disruption
Keywords: Fat Reduction; Lipolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XP1100RF group (Experimental): Subjects in the XP1100RF group will be treated with the XP1100RF device.
  Interventions: Device: XP1100RF

INTERVENTIONS:
Device: XP1100RF — Treatment of adipose tissue within the fat layer with XP1100RF device.

SUMMARY:
This study was designed to demonstrate safety and efficacy of the XP1100RF for non-invasive temporary reduction of thighs circumference by disruption of adipocyte cells.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open label study of thighs circumference reduction following 4 treatment sessions delivered once a week over a 4-week period. The objective of the study is to demonstrate the effectiveness of the treatment after 30-day in achieving thighs circumference reduction of ≥1 cm relative to the base line assessment.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 20 to 35 kg/m2.
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring and/or weight loss during study participation.
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting significant change in either direction during study participation.

Exclusion Criteria:

* Implanted electronic device such as a cardiac pacemaker, bladder stimulator, spinal cord stimulator or electrodes for a myoelectric prosthesis, etc.
* Diabetics dependent on insulin or oral hypoglycemic medications
* Known cardiovascular disease such as arrhythmias, congestive heart failure
* Cardiac surgeries such as cardiac bypass, heart transplant surgery, pacemakers.
* Prior surgical interventions for body sculpting of thighs such as liposuction
* Medical, physical or other contraindications for body sculpting/ weight loss
* Current use of medication known to affect weight levels and/or cause bloating or swelling and for which abstinence during the course of study participation is not safe or medically prudent
* Any medical condition known to affect weight levels and/or to cause bloating or swelling
* Active infection, wound or other external trauma to the area to be treated
* Pregnant, breast feeding, or planning pregnant before the end of the study
* Serious mental health illness
* Active or recurrent cancer or current chemotherapy and/or radiation treatment
* Negative affection to heat

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Thighs Circumference Reduction from Baseline at 30 days Follow Up | 30 days Follow Up
  The primary efficacy outcome measure is set to be a minimum of 80% of subjects at 30-day follow up evaluation to show thighs circumference reduction of ≥1 cm below the gluteal fold relative to the base line assessment.

SECONDARY OUTCOMES:
Adverse Events | 30 days Follow Up
  Absence of adverse events (AE) associated with the treatment procedure. Safety evaluations of skin reaction in the treatment area would be conducted at every treatment and follow up visits.
Adverse Events | 3 months Follow Up
  Absence of adverse events (AE) associated with the treatment procedure. Safety evaluations of skin reaction in the treatment area would be conducted at every treatment and follow up visits.
Subject satisfaction assessed by questionnaires | 30 days Follow Up
  Subject satisfaction as assessed by questionnaires administered at 30 days follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Radina Denkova, MD, Principal Investigator — Aesthe Beauty Clinic